CLINICAL TRIAL: NCT01982929
Title: An Evaluation of Post Caesarean-Section Pain Control Regimens: Non-Opioid Oral Regimen With and Without Transversus Abdominis Plane Block
Brief Title: Post Caesarean-Section Pain Control Regimens: Oral Regimen With and Without Transversus Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vicki Modest, MD (Other)
Responsible Party: Sponsor-Investigator, Vicki Modest, MD, Harvard Medical School Instructor in Clinical Anesthesia, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013P001906
Record Dates: First submitted 2013-10-28; First posted 2013-11-13 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Reduction in Post Ceasarean-section Related Pain in Study Group (TAP Block)
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham block & Oral Meds (Sham Comparator): Definition intervention. Sham procedure. Blocks mimicked the TAP blocks, but neither needle nor injectate was used. Patients had bilateral ultrasound scans over the lateral aspect of the abdomen. To mimic the injection of medicine, a blunt needleless syringe was firmly pressed on either side of the abdomen. An adhesive bandage was applied over the injection or sham injection sites.
  Interventions: Procedure: Sham block control
- TAP block & Oral Meds (Experimental): Definition intervention. TAP block (Bupivacaine 0.25% with epinephrine 1:400,000 50 cc). TAP blocks were placed using ultrasound-guided identification of the transversus abdominis fascial plane, and in-plane needle guidance. Injection sites were near the Triangle of Petit, located at the lateral edge of the mid-abdomen, near the iliac crests. After negative aspiration for blood, the local anesthetic was injected in 5 cc aliquots. The total dosage injected never exceeded 0.25 mg/kg of 0.25% bupivacaine with epinephrine 1:400,000.
  Interventions: Procedure: TAP block (Bupivacaine 0.25% with epinephrine)

INTERVENTIONS:
Procedure: TAP block (Bupivacaine 0.25% with epinephrine) — Ultrasound guided TAP blocks
  Arms: TAP block & Oral Meds
Procedure: Sham block control — A blunt needleless syringe was firmly pressed on either side of the abdomen.
  Arms: Sham block & Oral Meds

SUMMARY:
Patients at Mbarara Regional Referral Hospital (MRRH) in Uganda who present for routine caesarean sections often go without a set post-operative pain control regimen. Due to lack of established protocols and supplies of essential pain control medications are not reliable, upwards of 90% of women receive no postoperative pain control. There are regional techniques that are effective, easy to perform, low risk, and inexpensive. One of these techniques is a tranversus abdominis plane (TAP) block.

A TAP block is a regional anesthesia technique that provides analgesia to the parietal peritoneum as well as the skin and muscles of the anterior abdominal wall [1, 3-7]. First described just over a decade ago, it has undergone modifications in technique, and has been shown to be useful in providing 12-24 hours of significant post-operative pain relief for a wide array of surgical procedures [2]. It is best used as the cornerstone of a multi-modal approach to pain control and combines well with oral and intravenous opioid and non-opioid medications.

This is a technically straightforward procedure that involves injection of local anesthetic within the fascial plane located between the two deepest muscle layers (transversus abdominis and internal oblique muscles) of the lower abdominal wall. Given the simplicity of the TAP block and its long-lasting diminution in post-operative pain after many abdominal and pelvic surgeries, the incorporation of TAP blocks into post- caesarean section pain management should be considered as an achievable and simple remedy to the lack of reliable pain mediations after surgical delivery at MRRH.

This is a study that examines the efficacy of tranversus abdominis plane (TAP) blocks in providing post-operative analgesia after caesarean section under spinal anesthesia at Mbarara Regional Referral Hospital (MRRH) in Uganda, Africa. We will look at the value of TAP blocks in supplementing a routinely used (when available) post-operative non-opioid oral analgesic regimen.

Primary Hypothesis:

The administration of a TAP block on completion of caesarean section will decrease the level of pain as measured by a visual Numerical Rating Score (NRS) at 8, 16 and 24 hours, both at rest and with movement.

Secondary Hypotheses:

1. The administration of a TAP block on completion of caesarean section will increase the satisfaction score at 8, 16, and 24 hours; and
2. The administration of a TAP block will decrease or prevent the need for postoperative nurse- administered pethidine (meperidine) as a "rescue" medication.

This is a prospective, randomized, double-blind, sham controlled, single-center trial. A total of 240 patients will be enrolled in the study.

Following completion of the caesarean section, all patient will be screened for enrollment into the study. Enrollees will be randomly assigned to an arm via a predetermined undisclosed random number generator that will not be known by the staff at the MRRH. The anesthesiologist performing the TAP or sham block will be given a sealed envelope with the study arm which the patient has been randomized.

The study procedure is a TAP block and it will be placed on 50% of the enrollees.

TAP BLOCK:

Physicians who have been fully trained on the performance and potential risks of the technique will place TAP blocks under ultrasound-guidance. Briefly, under sterile conditions, ultrasound will be used to identify the targeted abdominal fascial plane. Once located, a predetermined amount of local anesthetic will be injected. This will be performed, bilaterally. The patient will be monitored during the block and for 30 minutes to follow.

SHAM BLOCK:

Sham blocks will consist of a non-invasive ultrasound scan over the abdomen. To mimic the injection of medicine, a dull/blunt object will be gently pressed on either side of the abdomen. The patient will be monitored during the sham block and for 30 minutes to follow.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the age of 18-44;
2. Greater than 50 kilograms in weight;
3. Status post a routine spinal anesthetic without sedation for an uncomplicated caesarean delivery via a low, transverse abdominal incision (Pfannenstiel);
4. In good health with no major medical problems including gastric ulcers, liver or renal dysfunction, and
5. Able to communicate freely with a provided non-family member interpreter fluent in the patient's language so that informed consent may be obtained.

Exclusion Criteria:

1. Patients with allergies to bupivicaine, paracetamol, or diclofenac;
2. Patients undergoing a surgical approach is other than a low, transverse abdominal incision (Pfannenstiel);
3. Pre-eclampsia, uterine rupture, placental abruption with this pregnancy;
4. Prior complicated abdominal surgery;
5. Medical history of gastric ulcers, liver or kidney dysfunction; and
6. Patient refusal to be involved in the study. -

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain level at rest, measured using the visual Numerical Rating Score (NRS) | NRS will be evaluated at T=0, 8, 16, and 24 hours after caesarean section.
  The NRS is an internationally accepted scale for measuring pain. It is a 0-10 whole interger scale where 0 is no pain and 10 is the worst. This study looks at the change in pain level over a 24 hour period.
Pain level with movement, measured using the visual Numerical Rating Score (NRS) | NRS will be evaluated at T=0, 8, 16, and 24 hours after caesarean section.
  The NRS is an internationally accepted scale for measuring pain. It is a 0-10 whole interger scale where 0 is no pain and 10 is the worst. This study looks at the change in pain level over a 24 hour period.

SECONDARY OUTCOMES:
Patient satisfaction with their pain control. The tool is an in person interview,with a yes/no answer | 24 hours post caesarean section

OTHER OUTCOMES:
Reduction in need for nurse-administered rescue pain medication over the 1st 24 hours post caesarean section as compared to control. This will be done by in person interview. | 24 hours post caesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda, Africa, Mbarara, Uganda

REFERENCES:
- [Background] Young MJ, Gorlin AW, Modest VE, Quraishi SA. Clinical implications of the transversus abdominis plane block in adults. Anesthesiol Res Pract. 2012;2012:731645. doi: 10.1155/2012/731645. Epub 2012 Jan 19. PMID 22312327